CLINICAL TRIAL: NCT06748755
Title: A Comparative Analysis of Ultrasound's Accuracy in Diagnosing Hepatocellular Carcinoma Using Histopathology as Gold Standard
Brief Title: A Comparative Analysis of Ultrasound's Accuracy in Diagnosing HC Using Histopathology as Gold Standard
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSAHS/Batch-Spring23/047
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Group 1 — To determine the sensitivity of ultrasound in detecting HCC

SUMMARY:
The study aims to evaluate the accuracy of ultrasound in diagnosing hepatocellular carcinoma (HCC), using histopathology as the gold standard. It addresses HCC's high global incidence and the utility of ultrasound as a non-invasive, cost-effective screening tool. Despite ultrasound's accessibility, its diagnostic limitations necessitate further investigation to improve clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Clinically suspected liver cancer patients undergoing ultrasound examination.
* Patients undergoing histopathological examination (liver biopsy or resection) for definitive diagnosis.

Exclusion Criteria:

- Patients with history of liver cancer treatment or inadequate data."

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: aim is to check the accuracy of Ultrasound's in Diagnosing Hepatocellular Carcinoma Using Histopathology as Gold Standard
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-02-20 (Estimated)

PRIMARY OUTCOMES:
ultrasound | 12 Months
  Sensitivity and Specificity analysis of Ultrasound as diagnostic tool, with histopathology as gold standard.

CONTACTS AND LOCATIONS:
Locations (1):
- Medcare International Hospital, Gujranwala, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No